CLINICAL TRIAL: NCT00518999
Title: Emotional and Cognitive Abilites of Schizophrenia Patients at Various Time Points
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Other Study IDs: 007-07-SHA
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Schizophrenia
Keywords: cognition, attention, memory, executive functions, illness-awareness, insight.
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Schizophrenia patients who performed earlier cognitive assessment as part of routine assessment for patients in the Shalvata Mental Health Center.

SUMMARY:
Longitudinal investigation of cognitive, emotional and illness awareness of schizophrenia outpatients (Shalvata Mental Health Center). The study uses computerized assessment of cognitive functioning and questionnaire to assess performance of patients assessed in the past as part of a routine clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Schizophrenia diagnosis by a senior psychiatrist (according to DSM-4 criteria).
2. Age between 18-65 (male and female).
3. Prior cognitive assessment in the Emotional-Cognitive Research Laboratory (Shalvata Mental Health Center)
4. Signed informed consent by participants.

Exclusion Criteria:

1. Hospitalization at the time of experiment.
2. A history of brain-injury or other neurological condition precluding participation in the study.
3. Guardianship.
4. Current alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-08; Study Completion 2008-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hilik Levkovitz, MD., Study Director — Shalvata Mental Health Center